CLINICAL TRIAL: NCT06564714
Title: Early Pharmacological Treatment of Acute Spasticity After Spinal Cord Injury to Promote Long-term Neurofunctional Recovery: a Randomized Clinical Trial
Brief Title: Early Pharmacological Treatment of Acute Spasticity After Spinal Cord Injury
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Andréane Richard-Denis, Principal investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-32-2023-2550
Record Dates: First submitted 2024-01-30; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Traumatic Spinal Cord Injury
Keywords: Trauma; Spinal Cord Injury; Baclofen; Spasticity
MeSH Terms: conditions — Wounds and Injuries; Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: 55 recruited participants will be randomized into the early baclofen treatment group or the control group.
Masking Description: Both investigators and trial participants will be fully aware of which treatment group the participants are in and what treatments are assigned to them.
  Participants will be randomized into the early baclofen treatment or control group using computer-generated random treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Baclofen treatment group (Experimental): Oral baclofen will be started as soon as any sign of acute spasticity consisting of spasms, velocity-dependent hypertonia and/or clonus is observed. Oral baclofen will be initiated the same day as when signs of spasticity are first observed.
  Dosage : oral administration of baclofen is started initially at 5 mg three times a day. The dose is increased every 7 days by 5 mg per intake (up to a maximum 80 mg total per day) until achieving an optimal response,
  Interventions: Drug: Early baclofen Intervention
- Control group (Other): The control group will receive the "usual routine care" as per which baclofen is prescribed only when acute spasticity becomes severe and problematic.
  In the presence of problematic spasticity, oral administration of baclofen is started initially at 5 mg three times a day. The dose is increased every 7 days by 5 mg per intake (up to a maximum 80 mg total per day) until achieving an optimal response.
  Interventions: Drug: Usual routine care

INTERVENTIONS:
Drug: Early baclofen Intervention — Baclofen is initiated as soon as any sign of acute spasticity.
  5 mg three times a day and is increased every 7 days by 5 mg per intake (up to a maximum 80 mg total per day) until achieving an optimal response, i.e. when spasticity is no longer problematic.
  Arms: Early Baclofen treatment group
Drug: Usual routine care — Baclofen is initiated only when acute spasticity is deemed problematic.
  5 mg three times a day and is increased every 7 days by 5 mg per intake (up to a maximum 80 mg total per day) until achieving an optimal response.
  Arms: Control group

SUMMARY:
The objective of this clinical trial is to evaluate if early detection of spasticity and immediate treatment with oral baclofen during acute care prevents problematic spasticity and improves neurofunctional recovery after tSCI.

The main questions it aims to answer are :

1. Assess the safety of early baclofen treatment during acute care after SCI.
2. Compare the neurofunctional outcomes between the early baclofen group and the control group up to 6 months after tSCI, in terms of mobility, global functional independence, neurological recovery, pain and spasticity.

The early baclofen group will receive oral administration of baclofen as soon as any sign of acute spasticity is observed. The dose is started initially at 5 mg three times a day and is increased every 7 days by 5 mg per intake (up to a maximum 80 mg total per day) until achieving an optimal response, i.e. when spasticity is no longer problematic. The control group however will receive the "usual routine care" at our institution as per which baclofen is initiated by the attending physician (i.e. physiatrist or spine surgeon) only when acute spasticity becomes severe and problematic.

DETAILED DESCRIPTION:
Spasticity is a condition in which muscles are abnormally stiff or tight, and interfere with normal movement. Following spinal cord injury (SCI), spasticity is common, affecting up to 70% of patients in the chronic stage 6 months or more after the injury. (1-4). After SCI, spasticity is due to a stretch reflex disorder of sensorimotor control following an upper motor neuron lesion, i.e. a lesion involving the neurons carrying the information within the spinal cord. Clinically, spasticity manifests as a complex syndrome of velocity-dependent hypertonia, clonus (rhythmic oscillating stretch reflex) and spasms (involuntary muscle contractions) that can have profound consequences on function and quality of life.

Traditionally, the clinical impact of spasticity has been mostly recognized during the subacute and chronic phases after SCI. Based upon the current management paradigm, the great majority of individuals with spasticity will receive pharmaceutical treatment for spasticity only during the rehabilitation period weeks or months after the injury when the clinical manifestations become severe and problematic. The investigators have challenged this long-held belief by proposing their paradigm shift towards early recognition and treatment of spasticity during the acute within the first month after SCI, after showing that about half of individuals will develop clinical signs of early spasticity during the acute hospitalization, and that acute spasticity is associated with poor long-term outcomes.

In particular, the investigators found that long-term mobility is significantly decreased in individuals presenting acute spasticity within the first month after the SCI. Our preliminary data suggest that prompt pharmacological treatment with baclofen - an anti-spasmodic medication - during the acute hospitalization improves neurological recovery in the presence of acute spasticity. Based on these preliminary findings, the overarching hypothesis of this study is that long-term neurofunctional outcomes are improved by early detection of acute spasticity and immediate treatment with oral baclofen.

Our team of experienced clinician-scientists specialized in SCI care therefore propose a single-site pilot randomized clinical trial including 55 patients admitted for a traumatic SCI (tSCI), in order to evaluate the safety and neurofunctional benefits of early baclofen treatment (i.e. as soon as any signs of spasticity are observed within the first month after the injury) during the acute hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Blunt (non-penetrating) traumatic SCI
* AIS grade A to D
* NLI between C0 and L1
* Patient willing and able to provide informed consent

Exclusion Criteria:

* Non-traumatic SCI (e.g. tumor, infection, transverse myelitis, etc.)
* AIS grade E upon admission
* Penetrating tSCI (from stab wound, gunshot injury, etc.)
* Cauda equina syndrome or NLI below L1
* Moderate or severe brain injury (mild traumatic brain injury not an exclusion criteria)
* Contraindication to oral baclofen use (needs clearance from attending physician and pharmacological consultant)
* Pre-existing neurological disorders (cerebrovascular disease, Parkinson's disease, multiple sclerosis, etc.)
* Major cognitive deficits precluding informed consent and/or assessments
* Unlikely to comply with scheduled visits (e.g. living in another country)
* Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Independence Measure (SCIM) | 6 months after the injury
  The primary outcome consists of the mobility subscore from the SCIM 6 months after the SCI with early baclofen treatment when compared to the control group.
  The SCIM will measure the ability of the 55 SCI patients to perform basic activities of daily living independently. There are 19 items divided into 3 subscales.
  A total score out of 100 is achieved, with the subscales weighted as follows:
  1. self-care: scored 0-20;
  2. respiration and sphincter management: scored 0-40; and
  3. mobility: scored 0-40
  Scores are higher in patients that require less assistance or fewer aids to complete basic activities of daily living and life support activities.
Adverse Events | From acute care to 6 months after the injury,
  Adverse events will be collected for both early baclofen treatment and control groups during acute care after SCI.

SECONDARY OUTCOMES:
Spastic reflexe assessment | All data on spastic reflexes will be collected from acute care to 6 months after the injury
  The Spinal Cord Assessment Tool for Spastic Reflexes (SCATS) will be used to measure spastic reflexes. This will be measured weekly, after hospital discharge and during outpatient follow-up visits 6 weeks and 6 months after the injury.
  The SCATS is split into 3 subscales, each addressing a seperate spasm.
  1) Clonus 2) Flexor spasms 3) Extensor spasms.
  For each subscale, the spasm is triggered and then rated. The degree of spasm is rated between 0 (no spasm) to 3 (severe spasm lasting longer than 10 seconds)
Muscle Spasticity assessment | All treatment and data on spasticity will be collected from acute care to 6 months after the injury.
  The Modified Ashworth Scale (MAS) will be used to measure spasticity for each muscle assessed.
  The MAS is a 6-point scale. Scores range from 0 (no increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension). This scale also adds a +1 scoring category to indicate resistance through less than half of the movement.
  Lower scores represent normal muscle tone and higher scores represent spasticity.
Spasticity frequency | All data on the frequency of spasticity will be collected from acute care to 6 months after the injury
  The Modified Penn Spasm Frequency Scale (mPSFS) will be used to quantify spasticity.
  It is a 2 component self-report measure in which the patients will report their perception of spasticity in regards to frequency and severity.
  The first component is a 5 point scale assessing the frequency with which spasms occur ranging from 0 (No spasms) to 4 (Spontaneous spasms occurring more than ten times per hour)
  The second component is a 3 point scale assessing the severity of spasms ranging from 1 (Mild) to 3 (Severe).
  The second component is not answered if the person indicates they have no spasms in part 1.
Spasticity impact | All data on the impact of spasticity will be collected from acute care to 6 months after the injury
  The Patient Reported Impact of Spasticity Measure (PRISM) measures the impact of SCI-related spasticity on quality of life from the patient's perspective.
  The PRISM consists of 41 items, divided into 7 subscales namely anxiety, psychological agitation, daily activities, assistance, positive impact, need for intervention, social embarrassment.
  It uses 5 point Likert Scale for scoring, 0 = Never true for me, 1 = Rarely true for me, 3 = Often true for me, 4 = Very often true for me. A higher score is considered unhealthy.
Neurological Assessment | From acute care to 6 months after the injury,
  The neurological status assessed from repeated neurological examinations between baseline and 6 months post-SCI will be measured using the International Standards for Neurological Classification of SCI (ISNCSCI)
  This impairment scale involves both a motor and sensory examination to determine the sensory and motor levels for the right and left side, the overall neurological level of the injury and completeness of the injury (i.e. whether the injury is complete or incomplete).
  Sensory evaluation is completed using a three-point scale for scoring. 0 = absent, 1 = altered (impaired or partial appreciation, including hyperesthesia), 2 = normal or intact (similar as on the cheek), NT = not testable.
  Motor evaluation is completed using a six-point scale for scoring ranging from 0 (total paralysis) to 5 (normal) active movement, full range of motion against gravity and full resistance in a muscle specific position expected from an otherwise unimpaired person)
Functional Assessment and Independent Walking | From acute care to 6 months after the injury,
  The 3rd version of the Spinal Cord Independence Measure (SCIM) will be used to report the ability of SCI patients to perform daily living activities independently,
  This questionnaire will measure Functional outcome of SCI partients before acute care and inpatient rehabilitation discharge, and at each follow-up visit.
Pain Assessment | From acute care to 6 months after the injury
  Pain assessment will be measured using the International Spinal Cord Injury Pain Basic Data Set (version 2.0).
  Information concerning pain's interference with physical and emotional function and sleep, probable pain diagnosis, pain location, pain intensity, and duration will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Andréane Richard-Denis, M.D., MSC, Principal Investigator — CIUSSS du Nord-de-l'île-de-Montréal-Hôpital du Sacré-Cœur de Montréal
Locations (1):
- CIUSSS du Nord-de-l'île-de-Montréal-Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cragg JJ, Tong B, Jutzeler CR, Warner FM, Cashman N, Geisler F, Kramer JLK. A Longitudinal Study of the Neurologic Safety of Acute Baclofen Use After Spinal Cord Injury. Neurotherapeutics. 2019 Jul;16(3):858-867. doi: 10.1007/s13311-019-00713-8. PMID 30725362
- [Background] Pandyan AD, Gregoric M, Barnes MP, Wood D, Van Wijck F, Burridge J, Hermens H, Johnson GR. Spasticity: clinical perceptions, neurological realities and meaningful measurement. Disabil Rehabil. 2005 Jan 7-21;27(1-2):2-6. doi: 10.1080/09638280400014576. No abstract available. PMID 15799140
- [Background] Adams MM, Hicks AL. Spasticity after spinal cord injury. Spinal Cord. 2005 Oct;43(10):577-86. doi: 10.1038/sj.sc.3101757. PMID 15838527
- [Background] Holtz KA, Lipson R, Noonan VK, Kwon BK, Mills PB. Prevalence and Effect of Problematic Spasticity After Traumatic Spinal Cord Injury. Arch Phys Med Rehabil. 2017 Jun;98(6):1132-1138. doi: 10.1016/j.apmr.2016.09.124. Epub 2016 Oct 22. PMID 27780743
- [Background] Ahuja CS, Wilson JR, Nori S, Kotter MRN, Druschel C, Curt A, Fehlings MG. Traumatic spinal cord injury. Nat Rev Dis Primers. 2017 Apr 27;3:17018. doi: 10.1038/nrdp.2017.18. PMID 28447605
- [Background] Ayoub S, Smith JG, Cary I, Dalton C, Pinto A, Ward C, Saverino A. The positive and the negative impacts of spasticity in patients with long-term neurological conditions: an observational study. Disabil Rehabil. 2021 Nov;43(23):3357-3364. doi: 10.1080/09638288.2020.1742803. Epub 2020 Mar 30. PMID 32223455
- [Background] Ehrmann C, Mahmoudi SM, Prodinger B, Kiekens C, Ertzgaard P. Impact of spasticity on functioning in spinal cord injury: an application of graphical modelling. J Rehabil Med. 2020 Mar 31;52(3):jrm00037. doi: 10.2340/16501977-2657. PMID 32103278
- [Background] D'Amico JM, Condliffe EG, Martins KJ, Bennett DJ, Gorassini MA. Recovery of neuronal and network excitability after spinal cord injury and implications for spasticity. Front Integr Neurosci. 2014 May 12;8:36. doi: 10.3389/fnint.2014.00036. eCollection 2014. PMID 24860447
- [Background] Bhimani RH, Anderson LC, Henly SJ, Stoddard SA. Clinical measurement of limb spasticity in adults: state of the science. J Neurosci Nurs. 2011 Apr;43(2):104-15. doi: 10.1097/jnn.0b013e31820b5f9f. PMID 21488584
- [Background] Adams MM, Ginis KA, Hicks AL. The spinal cord injury spasticity evaluation tool: development and evaluation. Arch Phys Med Rehabil. 2007 Sep;88(9):1185-92. doi: 10.1016/j.apmr.2007.06.012. PMID 17826466
- [Background] Lechner HE, Frotzler A, Eser P. Relationship between self- and clinically rated spasticity in spinal cord injury. Arch Phys Med Rehabil. 2006 Jan;87(1):15-9. doi: 10.1016/j.apmr.2005.07.312. PMID 16401432
- [Background] Levasseur A, Mac-Thiong JM, Richard-Denis A. Are early clinical manifestations of spasticity associated with long-term functional outcome following spinal cord injury? A retrospective study. Spinal Cord. 2021 Aug;59(8):910-916. doi: 10.1038/s41393-021-00661-1. Epub 2021 Jul 6. PMID 34230603
- [Background] Hiersemenzel LP, Curt A, Dietz V. From spinal shock to spasticity: neuronal adaptations to a spinal cord injury. Neurology. 2000 Apr 25;54(8):1574-82. doi: 10.1212/wnl.54.8.1574. PMID 10762496
- [Background] Dietz V, Sinkjaer T. Spastic movement disorder: impaired reflex function and altered muscle mechanics. Lancet Neurol. 2007 Aug;6(8):725-33. doi: 10.1016/S1474-4422(07)70193-X. PMID 17638613
- [Background] Li S, Francisco GE, Rymer WZ. A New Definition of Poststroke Spasticity and the Interference of Spasticity With Motor Recovery From Acute to Chronic Stages. Neurorehabil Neural Repair. 2021 Jul;35(7):601-610. doi: 10.1177/15459683211011214. Epub 2021 May 12. PMID 33978513